CLINICAL TRIAL: NCT06471530
Title: A Phase 1/2a, Open-label Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Effect on Body Weight of TE-8105 Administered Subcutaneously in Overweight/Obese Participants Without Diabetes
Brief Title: A Study to Investigate the Safety and Tolerability of TE-8105 in Overweight/Obese Participants Without Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immunwork, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TE-8105-101
Record Dates: First submitted 2024-06-06; First posted 2024-06-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A SAD Cohort 1 (Experimental): Each participant will receive TE-8105 administered by subcutaneous injection.
  Interventions: Drug: TE-8105 SAD Cohort 1
- Part A SAD Cohort 2 (Experimental): Each participant will receive TE-8105 administered by subcutaneous injection.
  Interventions: Drug: TE-8105 SAD Cohort 2
- Part A SAD Cohort 3 (Experimental): Each participant will receive TE-8105 administered by subcutaneous injection.
  Interventions: Drug: TE-8105 SAD Cohort 3
- Part A SAD Cohort 4 (Experimental): Each participant will receive TE-8105 administered by subcutaneous injection.
  Interventions: Drug: TE-8105 SAD Cohort 4
- Part A SAD Cohort 5 (Adaptive Cohort) (Experimental): Each participant will receive TE-8105 administered by subcuteneous injection.
  Interventions: Drug: TE-8105 SAD Cohort 5 (Adaptive cohort)
- Part B MAD Cohort 1 (Experimental): Each participant will receive TE-8105 administered by subcutaneous injection.
  Interventions: Drug: TE-8105 MAD Cohort 1
- Part B MAD Cohort 2 (Experimental): Each participant will receive TE-8105 administered by subcutaneous injection.
  Interventions: Drug: TE-8105 MAD Cohort 2

INTERVENTIONS:
Drug: TE-8105 SAD Cohort 1 — Each participant will receive one dose of TE-8105 0.5 up to 1.5mg injection via subcutaneous (SC) injection into the abdomen administered on Day 1.
  Arms: Part A SAD Cohort 1
Drug: TE-8105 SAD Cohort 3 — Each participant will receive one dose of TE-8105 1.5 mg or less than or equal to 2.5 mg injection via subcutaneous (SC) injection into the abdomen administered on Day 1.
  Arms: Part A SAD Cohort 3
Drug: TE-8105 SAD Cohort 5 (Adaptive cohort) — Each participant will receive one dose of TE-8105 less than or equal to 6 mg injection via subcutaneous (SC) injection into the abdomen administered on Day 1.
  Arms: Part A SAD Cohort 5 (Adaptive Cohort)
Drug: TE-8105 MAD Cohort 1 — Each participant will receive 0.5mg up to 1.5mg of TE-8105 injection via SC injection into the abdomen on Day 1 and then once every 2 weeks for 5 doses.
  Arms: Part B MAD Cohort 1
Drug: TE-8105 MAD Cohort 2 — Each participant will receive 9 doses of TE-8105 injection via SC injection into the abdomen starting from Day 1 every 2 weeks. Dose will be titrated up by 0.5mg every 4 weeks, with dose levels of 1.5mg (2 doses), 2.0 mg (2 doses), 2.5 mg (2 doses) and 3.0 mg (3 doses)
  Arms: Part B MAD Cohort 2
Drug: TE-8105 SAD Cohort 2 — Each participant will receive one dose of TE-8105 0.75mg injection via subcutaneous (SC) injection into the abdomen on Day 1.
  Arms: Part A SAD Cohort 2
Drug: TE-8105 SAD Cohort 4 — Each participant will receive one dose of TE-8105 3 mg or less than or equal to 5 mg injection via subcutaneous (SC) injection into the abdomen administered on Day 1.
  Arms: Part A SAD Cohort 4

SUMMARY:
This is a Phase 1/2a, first-in-human, prospective, open-label study to evaluate the safety, tolerability, PK, PD, and effect on body weight of TE-8105 in overweight/obese participants without diabetes. Study TE-8105-101 consists of 2 parts: Part A (single-ascending dose [SAD]) and Part B (multiple-ascending dose [MAD])

DETAILED DESCRIPTION:
Part A consists of 4 cohorts, with an optional adaptive cohort which may be opened if needed approximately 24 eligible participants will be assigned to Part A (SAD) (6 participants in each cohort). Part A is designed to evaluate the safety, tolerability, PK and effect on body weight of a single dose of 0.5 mg, 0.75 mg, 1.5 mg (or ≤ 2.5 mg), 3 mg (or ≤ 5 mg) TE-8105. Each participant will receive one dose of TE-8105 injection via subcutaneous (SC) injection into the abdomen administered on Day 1.

Part B consists of 2 cohorts. Approximately 14 participants will be assigned to Part B (MAD) (6 participants in B1 and 8 in B2 cohort). Part B is designed to evaluate the safety, tolerability, PK, PD, and effect on body weight of multiple SC doses 0.5 mg up to 3mg TE-8105 once every 2 weeks (Q2W). The dose levels and dosing interval of Part B may be adjusted based on the results of Part A. Each participant will receive 5 doses or 9 doses of TE-8105 injection via SC injection into the abdomen.

Progression from Part A to Part B will be based on the recommendation of the SRC.

ELIGIBILITY:
Inclusion Criteria:

Adults who are overweight or obese, do not have diabetes, and who are otherwise healthy, will be recruited. Main inclusion / exclusion criteria include but are not limited to:

* Male or female between 18 and 65 years old (both inclusive, at the time of informed consent).
* Have a BMI of ≥ 25 and ≤ 34.9 kg/m² or ≥ 23 and ≤ 32.5 kg/m² for Asian and Aboriginal participants.
* Have a stable body weight, defined as < 5% change in body weight, in either direction, during the Screening period (Day -28 to Day -1).
* Hemoglobin A1C (HbA1c) < 6.5%.
* Able and willing to provide written informed consent and any locally required authorization before performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria:

* Have attended any weight loss treatment or program (e.g., bariatric surgery, medication) within the 3 months prior to Screening, or have scheduled any weight loss treatment or program within the study period.
* Have had any exposure to GLP-1 analogs or other related compounds within the 3 months prior to Screening, or have a history of allergies to glucagon-like peptide-1 (GLP-1) analogs or related compounds.
* Have type 1 diabetes mellitus (T1DM) or type 2 diabetes mellitus (T2DM), a history of ketoacidosis, or hyperosmolar state/coma.
* Anything that the PI considers that would jeopardize the safety of the participant, or prevent complete participation in the study, or compromise the interpretation of study data.
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2.
* Have had a history of chronic pancreatitis or idiopathic acute pancreatitis.
* History of kidney dialysis or renal impairment measured as estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m² at Screening.
* Have GI disorder (for example, relevant esophageal reflux or gall bladder disease) or any GI disease that impacts gastric emptying (for example, gastric bypass surgery, pyloric stenosis, except appendectomy) or could be aggravated by GLP-1 analogs.
* Have obesity induced by other endocrinologic disorders (e.g., Cushing Syndrome) or diagnosed monogenetic or syndromic forms of obesity (e.g., Melanocortin 4 Receptor deficiency or Prader Willi Syndrome).
* Unwilling to refrain from commencing any new strenuous exercise programs (including weightlifting) from 7 days prior to admission to the study site until 28 days after the final dose.
* Women of childbearing potential (WOCBP) must be non-pregnant and must use an acceptable, highly effective double contraception from Screening until study completion.
* Males must use an acceptable, highly effective double contraception from Screening until study completion and must not donate sperm until at least 90 days after the last dose of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-06-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of TE-8105 by the incidence of treatment-related adverse events | SAD: From Screening until Day 43 (End of study) post dose. MAD: From Screening until Day 134 in Cohort B1 or Day 155 in Cohort B2 (End of study) post dose
Safety and tolerability of TE-8105 by the incidence of injection site reactions (ISRs) | SAD: On D 1, D 2, D 3, D 5, D 8. MAD Cohort B1: On D 1, D 2, D 3, D 8, D 15, D 29, D 43, D 57, D 64 post dose. MAD Cohort B2: On D 1, D2, D 3, D 5, D 8, D 15, D 29, D 43, D 57, D 71, D 85, D 99, D 113, D 117, D 120 and D 127
Number of participants with change in serum blood parameters | SAD: Scr, D-1, D2, D3, D8, D15, D29, D43 post dose. MAD B1: Scr, D-1, D2, D3, D8, D15, D29, D43, D57, D71, D92, D113, D134 post dose. MAD B2: Scr, D-1, D2, D3, D5, D8, D15, D29, D43, D57, D71, D85, D99, D113, D117, D120, D127, D141 and D155 post dose
  Laboratory assessment includes Hematology, coagulation and serum chemistry.
Number of participants with change in urine parameters | SAD: Scr, D-1, D2, D3, D8, D15, D29, D43 post dose. MAD B1: Scr, D-1, D2, D3, D8, D15, D29, D43, D57, D71, D92, D113, D134 post dose. MAD B2: Scr, D-1, D2, D3, D5, D8, D15, D29, D43, D57, D71, D85, D99, D113, D117, D120, D127, D141 and D155 post dose
  Laboratory assessment includes urinalysis
Number of participants with changes in the physical examination findings | Scr, D-1, D3, D8, D15 and D43 post dose. MAD B1: Scr, D-1, D3, D8, D15, D29, D43, D57, D71, D92, D113, D134 post dose. MAD B2: Scr, D-1, D2, D3, D5, D8, D15, D29, D43, D57, D71, D85, D99, D113, D117, D120, D127, D141 and D155 post dose
  Complete physical examinations include: general appearance, head, ears, eyes, nose, throat, neck (including thyroid and nodes), cardiovascular, respiratory, gastrointestinal, renal, neurological, musculoskeletal, skin, and other.
Number of participants with changes in 12 lead ECG findings | Scr, D-1, D1, D2, D3, D8, D15, D43 post dose. MAD B1: Scr, D-1, D1, D2, D3, D8, D15, D29, D43, D57, D71, D92, D113, D134 post dose. MAD B2: Scr, D-1, D2, D3, D5, D8, D15, D29, D43, D57, D71, D85, D99, D113, D117, D120, D127, D141 and D155 post dose
  ECG measurements to include Heart rate, PR, QRS, QT, and QTcF intervals.
Number of participants with changes in temperature | SAD: Scr, D-1, D1, D2, D3, D5, D8, D15, D43; MAD B1: Scr, D-1, D1, D2, D3, D8, D15, D29, D43, D57, D64, D71, D92, D113, D134; MAD B2: Scr, D-1, D2, D3, D5, D8, D15, D29, D43, D57, D71, D85, D99, D113, D117, D120, D127, D141 and D155 post dose
Number of participants with changes in blood pressure (BP) | SAD: Scr, D-1, D1, D2, D3, D5, D8, D15, D43; MAD B1: Scr, D-1, D1, D2, D3, D8, D15, D29, D43, D57, D64, D71, D92, D113, D134; MAD B2: Scr, D-1, D2, D3, D5, D8, D15, D29, D43, D57, D71, D85, D99, D113, D117, D120, D127, D141 and D155 post dose
  Systolic and diastolic BP will be measured
Number of participants with changes in heart rate (HR) | SAD: Scr, D-1, D1, D2, D3, D5, D8, D15, D43; MAD B1: Scr, D-1, D1, D2, D3, D8, D15, D29, D43, D57, D64, D71, D92, D113, D134; MAD B2: Scr, D-1, D2, D3, D5, D8, D15, D29, D43, D57, D71, D85, D99, D113, D117, D120, D127, D141 and D155 post dose
Number of participants with changes in respiratory rate (RR) | SAD: Scr, D-1, D1, D2, D3, D5, D8, D15, D43; MAD B1: Scr, D-1, D1, D2, D3, D8, D15, D29, D43, D57, D64, D71, D92, D113, D134; MAD B2: Scr, D-1, D2, D3, D5, D8, D15, D29, D43, D57, D71, D85, D99, D113, D117, D120, D127, D141 and D155 post dose

SECONDARY OUTCOMES:
PK Parameters : Maximum observed concentration (Cmax) | SAD: Predose and post dose on D1, D2, D3, D5, D8, D11, D15, D22, D29, D43 (EOS)
PK Parameters : Maximum observed concentration (Cmax) | MAD B1: Pre and post dose on D1, D2, D3, D8, D15, D29, D43, D57, D58, D59, D64, D71, D92, D113, D134; MAD B2: Pre and post dose on D1, D2, D3, D5, D8, D15, D29, D43, D57, D58, D71, D85, D99, D113, D114, D115, D117, D120, D127, D141 and D155
PK Parameters : Time to maximum observed concentration (Tmax) | SAD: Predose and post dose on D1, D2, D3, D5, D8, D11, D15, D22, D29, D43 (EOS)
PK Parameters : Time to maximum observed concentration (Tmax) | MAD B1: Pre and post dose on D1, D2, D3, D8, D15, D29, D43, D57, D58, D59, D64, D71, D92, D113, D134; MAD B2: Pre and post dose on D1, D2, D3, D5, D8, D15, D29, D43, D57, D58, D71, D85, D99, D113, D114, D115, D117, D120, D127, D141 and D155
PK Parameters : Area under the concentration-time curve (AUC) from time zero to the last measurable concentration (AUC 0-last) | SAD: Predose and post dose on D1, D2, D3, D5, D8, D11, D15, D22, D29, D43 (EOS)
PK Parameters : Area under the concentration-time curve (AUC) from time zero to the last measurable concentration (AUC 0-last) | MAD B1: Pre and post dose on D1, D2, D3, D8, D15, D29, D43, D57, D58, D59, D64, D71, D92, D113, D134; MAD B2: Pre and post dose on D1, D2, D3, D5, D8, D15, D29, D43, D57, D58, D71, D85, D99, D113, D114, D115, D117, D120, D127, D141 and D155
PK Parameters : Minimum observed concentration (Cmin) | MAD B1: Pre and post dose on D1, D2, D3, D8, D15, D29, D43, D57, D58, D59, D64, D71, D92, D113, D134; MAD B2: Pre and post dose on D1, D2, D3, D5, D8, D15, D29, D43, D57, D58, D71, D85, D99, D113, D114, D115, D117, D120, D127, D141 and D155
PK Parameters : AUC over a dosing interval (AUCτ). | MAD B1: Pre and post dose on D1, D2, D3, D8, D15, D29, D43, D57, D58, D59, D64, D71, D92, D113, D134; MAD B2: Pre and post dose on D1, D2, D3, D5, D8, D15, D29, D43, D57, D58, D71, D85, D99, D113, D114, D115, D117, D120, D127, D141 and D155
Number of participants with change in body weight from baseline with multiple doses of TE-8105. | Up to 20 weeks post first dose administration in MAD Cohort B1 and up to 23 weeks post first dose administration in MAD Cohort B2
Number of participants with change in Body mass index (BMI) from baseline with multiple doses of TE-8105. | Up to 20 weeks post first dose administration in MAD Cohort B1 and up to 23 weeks post first dose administration in MAD Cohort B2

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia